CLINICAL TRIAL: NCT00793910
Title: Oral Gabapentin Versus Placebo for Treatment of Postoperative Pain Following Photorefractive Keratectomy: A Randomized, Double-masked, Single Center, Placebo-controlled Clinical Trial
Brief Title: Oral Gabapentin Versus Placebo for Treatment of Postoperative Pain Following Photorefractive Keratectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Walter Reed Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Samantha B. Rodgers, MD, Assistant Director, Warfighter Refractive Eye Surgery Program and Research Center at Fort Belvoir, Fort Belvoir Community Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WRAMC WU# 08-6960
Record Dates: First submitted 2008-11-18; First posted 2008-11-19 (Estimated); Results first posted 2012-02-07 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Postoperative Pain
Keywords: Gabapentin; PRK; pain
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (2):
- Gabapentin (Active Comparator): oral medication
  Interventions: Drug: Gabapentin
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Gabapentin — Gabapentin 300 mg taken by mouth thrice daily for 7 days
  Arms: Gabapentin
Drug: placebo — placebo (sugar pill) taken by mouth thrice daily for 7 days
  Arms: placebo

SUMMARY:
The purpose of this study is to determine the effectiveness of an oral medication called gabapentin in reducing pain after Photorefractive Keratectomy (PRK) eye surgery and to assess the frequency of use of rescue medication interventions, defined as non-steroidal anti-inflammatory (NSAID) eye drops and oral narcotic medication.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and provide informed consent to participate in this study and complete follow-up visits.
* Planned Photorefractive keratectomy (PRK) at the WRAMC Center for Refractive Surgery.
* Male or female, of any race, and at least 21 years old at the time of the pre-operative examination, and have signed an informed consent. The lower age limit of 21 years is intended to ensure documentation of refractive stability.
* Access to transportation to meet follow-up requirements.

Exclusion Criteria:

* Any reason to be excluded for PRK.
* Female subjects who are pregnant, breast feeding or intend to become pregnant during the study. Female subjects will be given a urine pregnancy test prior to participating in the study to rule out pregnancy. [Pregnancy and breastfeeding are contraindications to refractive surgery in general, including PRK, whether participating in this study or not].
* Patients with known allergy, sensitivity or inappropriate responsiveness to Gabapentin or any of the medications used in the post-operative course.
* Patients with known depressed renal function.
* Any physical or mental impairment that would preclude participation in any of the examinations.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2008-07; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Walter Reed Army Medical Center, Washington D.C., District of Columbia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Gabapentin: Gabapentin 300mg taken by mouth thrice daily for 7 days
Period: Overall Study
Arm/Group | Gabapentin | Placebo
Started | 53 | 53
Completed | 48 | 46
Not Completed | 5 | 7
Not completed — discarded study pills | 0 | 1
Not completed — did not pick up medications | 1 | 1
Not completed — ineligible based on entry criteria | 2 | 3
Not completed — decided to undergo LASIK instead of PRK | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gabapentin | Placebo | Total
Number analyzed (Participants) | 48 | 46 | 94
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 48 | 46 | 94
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.7 (8) | 33.2 (7.9) | 31.9 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 42 | 39 | 81
Region of Enrollment [Number; unit: participants]
  United States | 48 | 46 | 94

OUTCOME MEASURES:

1. Primary Outcome: Level of Pain
Description: level of pain was measured using the Visual Analog Scale (VAS)ranging from 0 (none) to 10 (worst possible pain)
Time Frame: 2 hours postoperatively
Population: 11 patients who had alcohol-assisted PRK were removed from data analysis; 1 patient was disenrolled due to nausea secondary to oxycodone-acetaminophen (Percocet) intake
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 41 | 41
units on a scale | 3.85 (2.05) | 4.09 (2.38)

2. Secondary Outcome: Occurence of Use of Rescue Medication
Description: Occurrence of use of either ketorolac eyedrops(Acular) or oxycodone-acetaminophen tablet (Percocet), or both was measured
Time Frame: 2 hours to 4 days postoperatively
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: # of times rescue meds were used
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 41 | 41
# of times rescue meds were used | 7.54 (3.45) | 7.15 (3.9)

3. Primary Outcome: Level of Pain
Description: level of pain was measured using the Visual Analog Scale (VAS)ranging from 0 (none) to 10 (worst possible pain)
Time Frame: day 1 postoperatively
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 41 | 41
units on a scale | 3.00 (2.01) | 4.00 (1.97)

4. Primary Outcome: Level of Pain
Description: level of pain was measured using the Visual Analog Scale (VAS)ranging from 0 (none) to 10 (worst possible pain)
Time Frame: 3 days postoperatively
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 41 | 41
units on a scale | 2.09 (1.57) | 2.58 (2.08)

5. Primary Outcome: Level of Pain
Description: level of pain was measured using the Visual Analog Scale (VAS)ranging from 0 (none) to 10 (worst possible pain)
Time Frame: 4 days postoperatively
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 41 | 41
units on a scale | 1.30 (1.16) | 1.86 (1.96)

ADVERSE EVENTS:
Arm/Group | Gabapentin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/53
Other Adverse Events (participants affected / at risk) | 0/53 | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All materials that reflects the WRAMC affiliation must be approved and properly cleared before the material is submitted for public dissemination and publication. All publications whereby WRAMC is cited in the bylines will state on the cover page the following sample disclaimer: "The views expressed in this [article, book chapter, speech, presentation, etc.] are those of the author(s) and do not reflect the official policy of the Department of Army, Department of Defense, or U.S. Government."